CLINICAL TRIAL: NCT05324449
Title: Epidiolex® For The Treatment Of Anxiety Comorbidity in Refractory Pediatric Epilepsy
Brief Title: Epidiolex® for Anxiety in Pediatric Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Jay Salpekar, M.D., Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00282248
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Epilepsy
MeSH Terms: conditions — Anxiety Disorders; Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Other): open label treatment intervention
  Interventions: Drug: Cannabidiol 100 MG/ML

INTERVENTIONS:
Drug: Cannabidiol 100 MG/ML — pharmaceutical grade cannabidiol
  Other Names: Epidiolex

SUMMARY:
This is a prospective open label study assessing the efficacy and tolerability of pharmaceutical grade cannabidiol--Epidiolex (R), for the treatment of anxiety in pediatric patients with pediatric epilepsy that has been difficult to treat and requires ongoing use of anticonvulsant medication.

DETAILED DESCRIPTION:
This study is an open label, adjunctive, proof of concept clinical trial. Prospective participants will be considered for the study if neurologic status suggests the need for continued treatment, and behavioral characteristics are clinically significant. All participants will receive active treatment, involving flexible dose titration of Epidiolex® and will be monitored for a period of four months. The study will be monitored and overseen by the Johns Hopkins Hospital Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of epilepsy, characterized by focal or generalized seizures. All participants will have active epilepsy that requires treatment with anticonvulsant medication.
2. No episodes of seizure clusters of status epilepticus within 30 days prior to entry into the study.
3. Established symptoms of anxiety with functional impairment.
4. Baseline behavioral criteria for inclusion will include subscale scores for anxiety above the norm for age and gender inth e 60 days prior to the study on one of the following:
5. Male or female participants equal to or above age 6 and below age 18 at the start of the study. No exclusion will be made on the basis of gender or minority status.
6. Ability to administer medicine orally
7. Previous subjects who failed at any point to meet continuation criteria and withdrew early may be considered for re-enrollment by the PI on a case-by-case basis.
8. Participant or legal caregiver capable of providing informed consent and fully capable of monitoring the subject's disease process and compliance with treatment.
9. Participants who are sexually active, must agree to sexual abstinence, or, to use an approved birth control method for the full duration of study participation.
10. No active use of CBD products within the 14 days prior to screening visit and commitment to only use study product for the duration of the study.

Exclusion Criteria:

1. Baseline lab tests for liver specific transaminase, ALT, over the upper limit of normal (ULN).
2. Previous allergic or hypersensitivity reactions to Epidiolex® or cannabidiol
3. No access to a phone or internet to complete remote visits (in-person visits acceptable for participants without devices)
4. Active substance abuse or dependence
5. Presence of psychotic illness or imminent risk of harm to self or others.
6. Current standing use of benzodiazepines (except as "rescue" medicine)
7. Serious unstable medical or neurologic conditions such as HIV, liver or kidney disease, cancer or diabetes.
8. Presence of Epilepsy Syndrome such as Sturge-Weber Syndrome that will be more suitable as a candidate in alternate research studies.
9. Participation in a previous experimental drug study within 30 days of baseline visit.
10. Cognitive functional capacity or English literacy that is insufficient to assure validity of clinical rating scales
11. Insufficient capacity of caregiver or legal guardian to understand and appropriately consent for study procedures
12. No exclusions for existing AEDs will be absolute, though consideration of additional monitoring will be in place for patients taking clobazam or valproate.
13. Pregnant, planning to become pregnant, breast feeding, or failing to use an appropriate method of contraception.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
CGI-I | 16 weeks
  Mean of Clinical Global Impression-Improvement (CGI-I) from baseline. The CGI is rated on a 7-point scale. (lower score represents a better outcome: 1/ High score represents minimum improvement: 7)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Salpekar, Principal Investigator — Principal Investigator
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
data will be assembled and de-identified and analyzed in aggregate

REFERENCES:
- [Background] Abu-Sawwa R, Scutt B, Park Y. Emerging Use of Epidiolex (Cannabidiol) in Epilepsy. J Pediatr Pharmacol Ther. 2020;25(6):485-499. doi: 10.5863/1551-6776-25.6.485. PMID 32839652